CLINICAL TRIAL: NCT05678023
Title: Multicentre Randomized Trial on the Timing and Effect of Contrast Media on Patients with Adhesive Small Bowel Obstruction
Brief Title: Study About Contrast Media
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Collaborators: North Estonia Medical Centre (Other)
Responsible Party: Principal Investigator, Liis Jaanimäe, General Surgeon, PhD student, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22031
Record Dates: First submitted 2022-12-04; First posted 2023-01-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sealed envelope randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contrast media 4 hours (Active Comparator): Patients will receive contrast media after 4 hours of nasogastric decompression
  Interventions: Other: Effect on contrast media depending on the time of its administratsion
- Contrast media 24 hours (Active Comparator): Patients will receive contrast media after 24 hours of nasogastric decompression
  Interventions: Other: Effect on contrast media depending on the time of its administratsion

INTERVENTIONS:
Other: Effect on contrast media depending on the time of its administratsion — CM is a common practice when it comes to the management of small bowel obstruction. However there is no consensus as when it should be administered

SUMMARY:
Patients hospitalized with adhesive small bowel obstruction (SBO) are randomized to 2 study groups at admission after signing an informed consent form. Water-soluble contrast media (CM) will be administered after 4 or after 24 hours of nasogastric- tube decompression.

DETAILED DESCRIPTION:
Patients presenting with symptoms of small bowel obstruction (SBO) will be evaluated and if the diagnosis of adhesive small bowel obstruction is made it must be decided what is the treatment of choice.

If immediate surgery is needed- it will not be delayed If patients are eligible for conservative management- they will be randomized to 2 study groups- contrast media (CM) after 4 hours of nasogastric-tube decompression and after 24 hours of nasogastric-tube decompression.

Contrast media challenge acquires radiographs (X-rays) to be taken after an interval (common practice) decided by the surgeon.

If at any point patient needs surgery- it will not be delayed. The results are compared. The hypothesis is, that if CM is administered sooner- it will help SBO resolution

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Adhesive small bowel obstruction diagnosed (clinical, laboratory and radiologic evaluation
* No peritonitis present, no need for an emergent surgery
* Patients sign an informed consent

Exclusion Criteria:

* Patients younger than 18 yeas
* Patients with mechanical small bowel obstruction caused by incarcerated hernias
* Patients with mechanical small bowel obstruction caused by carcinomatosis
* Patients with paralytic small bowel obstruction
* Patients who have undergone surgery within 6 weeks
* Patients who do not want to be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
SBO resolution | Period of hospitalization- approximately 5 days
  SBO resolution with conservative measures
  * passing gas
  * bowel movement
  * CM in the colon on the X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Liis Jaanimäe, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided